CLINICAL TRIAL: NCT04941729
Title: A Prospective, Multi-center, Randomized, Controlled Study to Evaluate the Safety and Efficacy of the OR3O™ Dual Mobility System Versus Conventional Single Bearing Design Total Hip System in Primary Total Hip Arthroplasty (THA) Procedures.
Brief Title: Study to Evaluate the Safety and Efficacy of OR3O™ Dual Mobility System vs. Conventional Single Bearing Design Total Hip System
Acronym: OR3O
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change on clinical and marketing strategy for the devices
Sponsor: Smith & Nephew Medical (Shanghai) Ltd (Industry)
Responsible Party: Sponsor
Organization: Smith & Nephew, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OR3O.2019.10 (CHINA)
Record Dates: First submitted 2021-05-13; First posted 2021-06-28 (Actual); Results first posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2024-11

CONDITIONS: Degenerative Hip Joint Disease; Rheumatoid Arthritis (RA); Femoral Neck Fractures; Avascular Necrosis of Femoral Head; Osteoarthritis (OA); Hip Dislocation; Hip Fractures
Keywords: Total Hip Arthroplasty (THA)
MeSH Terms: conditions — Osteoarthritis, Hip; Arthritis, Rheumatoid; Femoral Neck Fractures; Femur Head Necrosis; Osteoarthritis; Hip Dislocation; Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Arm (dual mobility) (Experimental): OR3O™ Dual Mobility in subjects who undergo Primary THA.
  Interventions: Device: OR3O™ - Dual Mobility System
- Controlled Arm (conventional) (Active Comparator): A conventional, single-bearing design Total Hip System in subjects who undergo Primary THA.
  Interventions: Device: Conventional

INTERVENTIONS:
Device: OR3O™ - Dual Mobility System — OR3O™ Dual Mobility System is comprised of a diffusion-hardened, oxidized zirconium acetabular liner (OR3O™ Liner), and an insert of highly cross-linked polyethylene (OR3O™ XLPE Insert).
  Arms: Study Arm (dual mobility)
Device: Conventional — A conventional, single-bearing design Total Hip System comprised of R3™ Acetabular Shell with XLPE liner and a Smith & Nephew Oxinium (Ox) femoral head.
  Arms: Controlled Arm (conventional)

SUMMARY:
The purpose of this study is to compare OR3O™ Dual Mobility System to a conventional, single-bearing design Total Hip System in subjects who undergo Primary THA. Data collected in this study will be used to support National Medical Products Administration (NMPA) regulatory approval of OR3O™ Dual Mobility System in China as well as to support and maintain product registration in global markets.

Primary Objective: Assess safety and efficacy of the OR3O™ Dual Mobility System in Primary THA at 1 year postoperative.

Secondary Objective(s): Assess safety and efficacy of the OR3O™ Dual Mobility System and compatible components in Primary THA up to 2 years after surgery.

Other Objective(s): Assess the hip dislocation and hospital readmission up to 2 years after device implantation.

4 study sites in China.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a suitable candidate for implanting the OR3O™ Dual Mobility System or single-bearing design Total Hip System in primary total hip replacement in the Investigator's judgement.
* Subject is skeletally mature in the Investigator's judgement.
* Subject is 18 - 80 years old (inclusive).
* Subject is receiving total hip replacement for the first time on the affected hip.
* Subject has any of the following conditions:

  * Advanced degeneration of the hip joint as a result of degenerative, post-traumatic, or rheumatoid arthritis(RA);
  * Fracture or avascular necrosis of the femoral head;
  * All forms of osteoarthritis(OA);
  * Patients with hips at risk of dislocation;
  * Femoral neck fracture or proximal hip joint fracture.
* Subject provides written informed consent for study participation using an Ethical Committee (EC) approved consent form before any study procedures are performed, including pre-operative data review and/or collection of data on electronic Case Report Forms (eCRFs).
* Subject is willing and able to participate in required follow-up visits and is able to complete study activities.
* Subjects with preoperative HHS ≤ 79 (fair or worse category).

Exclusion Criteria:

* Subject has conditions that would eliminate or tend to eliminate adequate implant support or prevent the use of an appropriately-sized implant, e.g.:

  * blood supply limitations;
  * insufficient quantity or quality of bone support, e.g., osteoporosis, metabolic disorders which may impair bone formation, radioactive bone disease, tumor around hip joint, and osteomalacia;
  * infections or other conditions which may lead to increased bone resorption.
* Subject has dysplasia of hip joint with CROWE Grade III, IV.
* Subject has weak constitution or failing to endure the surgery due to other diseases of the body.
* Subject has bodily disease(s) that may interfere with THA survival or outcome.
* Subject has life expectancy of less than 2 years.
* Subject has mental or neurological conditions which impair the subject's ability or willingness to restrict activities that may put the affected limb at risk.
* Subject has physical conditions or activities which tend to place extreme loads on implants, e.g., Charcot joints, muscle deficiencies, multiple joint disabilities.
* Subject has neuromuscular dysfunctions (paralysis, myolysis and abductor muscle weakness) which will cause unstable hip joint or abnormal gait after surgery.
* Subject has a mental or neurological condition that would pre-empt their ability or willingness to participate in the study including mental illness, mental retardation, drug or alcohol abuse.
* Subject has an active infection - systemic or at the site of intended surgery.
* Subject has a Body Mass Index ≥ 40.0 kg/m².
* Subject has a known allergy to any component of the devices used in the study.
* Subject is pregnant or breast feeding.
* Subject is entered in another investigational drug, biologic, or device study within 30 days of active study participation.
* Subjects that are expected with poor compliance.
* Subjects with complications of other diseases are limited to participate in the research, not able to comply with the follow-up or have impact on scientific integrity.
* Subjects with preoperative HHS ≥ 80 (good to excellent category).
* Subject has other diseases or conditions that investigator considers not appropriate to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-06-24 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2023-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Li Cao, Principal Investigator — First Affiliated Hospital of Xinjiang Medical University
Locations (4):
- China (4):
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Peking University Third Hospital, Beijing
  - The Ninth People's Hospital affiliated to Shanghai Jiao Tong University Medical College, Shanghai
  - The First Affiliated Hospital of Xinjiang Medical University, Xinjiang

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 24 participants were consented. Two participants were excluded from the study prior to receiving study treatment due to screen failure and withdrawal by the participant.
Period: Overall Study
Arm/Group | Study Arm (Dual Mobility) | Controlled Arm (Conventional)
Started | 11 | 11
Completed | 0 | 0
Not Completed | 11 | 11
Not completed — Death | 0 | 1
Not completed — Study terminated by sponsor | 11 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Arm (Dual Mobility) | Controlled Arm (Conventional) | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (10.5) | 65.1 (9.6) | 60.8 (10.8)
Age, Customized [Count of Participants; unit: Participants]
  Age Category: < 60 years | 8 | 2 | 10
  Age Category: ≥ 60 years | 3 | 9 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 9 | 12
  Male | 8 | 2 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Chinese | 11 | 11 | 22
  Race: Han | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 11 | 11 | 22
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.2 (3.3) | 23.5 (3.7) | 24.4 (3.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Excellent or Good Harris Hip Score (HHS) at 12 Months
Description: Number of participants with an excellent (≥ 90) or good (80-89) Harris Hip Score at 12 months postoperative (No/Yes).
  The Harris Hip Score is a joint specific score that consists of 10 items covering domains of pain (1 item, 0-44 points), function (7 items, 0-47 points), functional activities, absence of deformity (1 item, 0 or 4 points), and hip range of motion (2 items, 0-5 points). Scores range from 0 (worst) to 100 (best).
Time Frame: 12 months
Population: Safety Analysis (SAF) population included participants assigned to a study arm with data collected for the outcome and time frame specified.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Arm (Dual Mobility) | Controlled Arm (Conventional)
Number analyzed (Participants) | 7 | 7
Participants
  No | 1 | 4
  Yes | 6 | 3

2. Secondary Outcome: Survivorship of the OR3O™ Dual Mobility System
Description: Survivorship of the OR3O™ Dual Mobility System measured by Kaplan-Meier survival estimate. Survivorship was defined as number of hips with no revision due to any reason.
Time Frame: 6 weeks, 3 months, 6 months, and 12 months
Population: Safety Analysis (SAF) population included participants assigned to a study arm with data collected for the outcome and time frame specified. Data was only collected up to the 12 month time point due to premature termination of the study.
Measure: Count of Units; unit: hips
Units Other Than Participants: hips
Arm/Group | Study Arm (Dual Mobility) | Controlled Arm (Conventional)
Number analyzed (Participants) | 11 | 11
Number analyzed (hips) | 11 | 11
hips
  6 weeks | 11 | 11
  3 months: number analyzed (Participants) | 10 | 10
  3 months: number analyzed (hips) | 10 | 10
  3 months | 10 | 10
  6 months: number analyzed (Participants) | 10 | 9
  6 months: number analyzed (hips) | 10 | 9
  6 months | 10 | 9
  12 months: number analyzed (Participants) | 5 | 5
  12 months: number analyzed (hips) | 5 | 5
  12 months | 5 | 5

3. Secondary Outcome: Harris Hip Score (HHS)
Description: The Harris Hip Score is a joint specific score that consists of 10 items covering domains of pain, function, functional activities, absence of deformity, and hip range of motion. Scores range from 0 (worst) to 100 (best).
Time Frame: Preoperative, 6 weeks, 6 months, and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Arm (Dual Mobility) | Controlled Arm (Conventional)
Number analyzed (Participants) | 11 | 11
score on a scale
  Preoperative | 34.09 (22.42) | 31.55 (19.44)
  6 weeks: number analyzed (Participants) | 1 | 1
  6 weeks | 71 (NA) — Standard Deviation could not be calculated because data was only collected for one participant | 51 (NA) — Standard Deviation could not be calculated because data was only collected for one participant
  6 months: number analyzed (Participants) | 10 | 9
  6 months | 73.1 (7.45) | 72.33 (6.78)
  12 months: number analyzed (Participants) | 7 | 7
  12 months | 81.86 (4.74) | 75.71 (8.65)

4. Secondary Outcome: EuroQol (European Quality of Life) Five-dimensional Five-level (EQ-5D-5L) Score: Visal Analogue Scale (VAS) Score
Description: The EQ-5D-5L is composed of the EQ-5D-5L descriptive system and the EQ Visual Analogue scale (EQ VAS). The EQ VAS score is on a scale of 0 to 100 with 0 indicating 'the worst health you can imagine' and 100 indicating 'the best health you can imagine' (i.e., a higher score is a better outcome).
Time Frame: Preoperative, 6 weeks, 6 months, and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Arm (Dual Mobility) | Controlled Arm (Conventional)
Number analyzed (Participants) | 11 | 11
score on a scale
  Preoperative | 51.82 (27.14) | 55.91 (17.44)
  6 weeks: number analyzed (Participants) | 2 | 1
  6 weeks | 72.5 (3.54) | 80 (NA) — Standard Deviation could not be calculated because data was only collected for one participant
  6 months: number analyzed (Participants) | 10 | 9
  6 months | 78 (11.35) | 76.67 (9.68)
  12 months: number analyzed (Participants) | 7 | 7
  12 months | 81.43 (9.00) | 79.29 (8.86)

5. Secondary Outcome: EuroQol (European Quality of Life) Five-dimensional Five-level (EQ-5D-5L) Score: Health Score
Description: The EQ-5D-5L is composed of the EQ-5D-5L descriptive system and the EQ Visual Analogue scale (EQ VAS). The descriptive system comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression) to create a combined Health Score. The combined Health Score is on a scale of 0 to 1 with a higher score indicating a better outcome.
Time Frame: Preoperative, 6 weeks, 6 months, and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Arm (Dual Mobility) | Controlled Arm (Conventional)
Number analyzed (Participants) | 11 | 11
score on a scale
  Preoperative | 0.36 (0.30) | 0.37 (0.25)
  6 weeks: number analyzed (Participants) | 2 | 1
  6 weeks | 0.63 (0.02) | 0.69 (NA) — Standard Deviation could not be calculated because data was only collected for one participant
  6 months: number analyzed (Participants) | 10 | 9
  6 months | 0.74 (0.11) | 0.71 (0.14)
  12 months: number analyzed (Participants) | 7 | 7
  12 months | 0.79 (0.11) | 0.73 (0.19)

6. Secondary Outcome: Hip Disability and Osteoarthritis Outcome Score for Joint Replacement (HOOS JR.)
Description: The HOOS JR. is a short-form survey based on the Hip Disability and Osteoarthritis Outcome Score (HOOS) that specifically focuses on the outcome after Total Hip Arthroplasty (THA). HOOS JR. accesses pain and joint awareness during the activities of daily living. The scores range from 0 to 100 with 0 indicating total hip disability (i.e., the worst outcome) and 100 indicating perfect hip health (i.e., the best outcome).
Time Frame: Preoperative, 6 weeks, 6 months, and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Study Arm (Dual Mobility) | Controlled Arm (Conventional)
Number analyzed (Participants) | 11 | 11
score on a scale
  Preoperative | 54.29 (23.57) | 46.69 (18.37)
  6 weeks: number analyzed (Participants) | 2 | 1
  6 weeks | 64.68 (8.13) | 67.52 (NA) — Standard Deviation could not be calculated because data was only collected for one participant
  6 months: number analyzed (Participants) | 10 | 9
  6 months | 80.42 (8.88) | 79.25 (15.29)
  12 months: number analyzed (Participants) | 7 | 7
  12 months | 83.83 (10.14) | 74.91 (15.12)

7. Secondary Outcome: Radiographic Assessment - Implant Position/Orientation
Description: Implant position/orientation determined by acetabular cup position from radiographs performed with the participant in a supine position. Participant implant position was categorized as one of the following:
  * Unchanged
  * Varus tilted
  * Valgus tilted
  * Subsidence
Time Frame: 6 months and 12 months
Population: Safety Analysis (SAF) population included participants assigned to a study arm with data collected for the outcome and time frame specified. Data was only collected up to the 12 month time point due to premature termination of the study. Radiographs only collected at 6 months & 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Arm (Dual Mobility) | Controlled Arm (Conventional)
Number analyzed (Participants) | 7 | 7
Participants
  6 months: number analyzed (Participants) | 4 | 3
  6 months: Unchanged | 4 | 3
  6 months: Varus tilted | 0 | 0
  6 months: Valgus tilted | 0 | 0
  6 months: Subsidence | 0 | 0
  12 months: Unchanged | 7 | 7
  12 months: Varus tilted | 0 | 0
  12 months: Valgus tilted | 0 | 0
  12 months: Subsidence | 0 | 0

8. Secondary Outcome: Radiographic Assessment - Implant Subsidence/Migration
Description: Acetabular Cup Migration was determined based on cup fixation from radiographs with the subject in a supine position. Participant implant subsidence/migration was categorized as one of the following:
  * Unchanged
  * Migration cranial
  * Migration medial
  * Tilted
Time Frame: 6 months and 12 months
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Study Arm (Dual Mobility) | Controlled Arm (Conventional)
Number analyzed (Participants) | 7 | 7
Participants
  6 months: number analyzed (Participants) | 4 | 3
  6 months: Unchanged | 4 | 3
  6 months: Migration cranial | 0 | 0
  6 months: Migation medial | 0 | 0
  6 months: Tilted | 0 | 0
  12 months: Unchanged | 7 | 7
  12 months: Migration cranial | 0 | 0
  12 months: Migation medial | 0 | 0
  12 months: Tilted | 0 | 0

9. Secondary Outcome: Radiographic Assessment - Heterotopic Ossification
Description: Heterotopic Ossification determined from radiographs performed with the subject in a supine position using Brooker Classification. Heterotopic ossification for the participant was classified as one of following:
  * Grade 0 (None, no islands of bone)
  * Grade I (Islands of bone within the soft tissues about the hip)
  * Grade II (Bone spurs from the pelvis or proximal end of the femur, leaving at least 1 cm between opposing bone surfaces)
  * Grade III (Bone spurs from the pelvis or proximal end of the femur, reducing the space between opposing bone surfaces to less than 1 cm)
  * Grade IV (Apparent bone ankylosis of the hip)
Time Frame: 6 months and 12 months
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Study Arm (Dual Mobility) | Controlled Arm (Conventional)
Number analyzed (Participants) | 7 | 7
Participants
  6 months: number analyzed (Participants) | 4 | 3
  6 months: Grade 0 | 4 | 3
  6 months: Grade I | 0 | 0
  6 months: Grade II | 0 | 0
  6 months: Grade III | 0 | 0
  6 months: Grade IV | 0 | 0
  12 months: Grade 0 | 7 | 7
  12 months: Grade I | 0 | 0
  12 months: Grade II | 0 | 0
  12 months: Grade III | 0 | 0
  12 months: Grade IV | 0 | 0

10. Secondary Outcome: Radiographic Assessment - Radiolucencies
Description: Radiolucencies in the Acetabular Cup are defined as the presence of a linear gap or "halo" along the acetabular bone-implant interface identified from radiographs performed with the subject in a supine position. The presence of radiolucent lines for participants in any cup zones were categorized as either 'Yes' or 'No'.
Time Frame: 6 months and 12 months
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Study Arm (Dual Mobility) | Controlled Arm (Conventional)
Number analyzed (Participants) | 7 | 7
Participants
  6 months: number analyzed (Participants) | 4 | 3
  6 months: Yes | 0 | 0
  6 months: No | 4 | 3
  12 months: Yes | 0 | 0
  12 months: No | 7 | 7

11. Secondary Outcome: Radiographic Assessment - Osteolysis
Description: Osteolysis was determined from radiographs performed with the subject in a supine position. The presence of osteolysis in any cup zones for the participant identified as 'Yes' or 'No'. Presence of osteolysis indicated a ballooning / scalloping, progressive, periacetabular, bony destructive lesion with a maximum dimension > 5 millimeters (mm).
Time Frame: 6 months and 12 months
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Study Arm (Dual Mobility) | Controlled Arm (Conventional)
Number analyzed (Participants) | 7 | 7
Participants
  6 months: number analyzed (Participants) | 4 | 3
  6 months: Yes | 0 | 0
  6 months: No | 4 | 3
  12 months: Yes | 0 | 0
  12 months: No | 7 | 7

12. Secondary Outcome: Radiographic Assessment - Implant Loosening
Description: Implant loosening was determined from radiographs performed with the subject in a supine position. The presence of loosening indicated apparent imaging features of loosening at the acetabular bone-implant interface including significant radiolucency or change in position of the acetabular cup indicating a loss of fixation. Implant loosening based on stem fixation for cemented stems for the participant was categorized as one of the following:
  * Not applicable
  * No loosening
  * Possible loosening
  * Probable loosening
  * Definite loosening
Time Frame: 6 months and 12 months
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Study Arm (Dual Mobility) | Controlled Arm (Conventional)
Number analyzed (Participants) | 7 | 7
Participants
  6 months: number analyzed (Participants) | 4 | 3
  6 months: Not applicable | 0 | 0
  6 months: No loosening | 4 | 3
  6 months: Possible loosening | 0 | 0
  6 months: Probable loosening | 0 | 0
  6 months: Definite loosening | 0 | 0
  12 months: Not applicable | 0 | 0
  12 months: No loosening | 7 | 7
  12 months: Possible loosening | 0 | 0
  12 months: Probable loosening | 0 | 0
  12 months: Definite loosening | 0 | 0

13. Secondary Outcome: Radiographic Assessment - Stress Shielding
Description: Image review by investigator of radiographs performed with the subject in a supine position to identify presence of medial stress shielding. Stress shielding for the participant based on the presence (Yes/No) of the following:
  * Atrophy in any Cup Zones
  * Atrophy in any Stem Zones
Time Frame: 6 months and 12 months
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Study Arm (Dual Mobility) | Controlled Arm (Conventional)
Number analyzed (Participants) | 7 | 7
Participants
  6 months: Atrophy in any Cup Zones: number analyzed (Participants) | 4 | 3
  6 months: Atrophy in any Cup Zones: Yes | 0 | 0
  6 months: Atrophy in any Cup Zones: No | 4 | 3
  6 months: Atrophy in any Stem Zones: number analyzed (Participants) | 4 | 3
  6 months: Atrophy in any Stem Zones: Yes | 0 | 0
  6 months: Atrophy in any Stem Zones: No | 4 | 3
  12 months: Atrophy in any Cup Zones: Yes | 0 | 0
  12 months: Atrophy in any Cup Zones: No | 7 | 7
  12 months: Atrophy in any Stem Zones: Yes | 0 | 0
  12 months: Atrophy in any Stem Zones: No | 7 | 7

14. Secondary Outcome: Radiographic Assessment - Periprosthetic Fractures
Description: Image review by investigator to identify presence of periprosthetic fractures (yes/no). An AP and a lateral view radiograph are required to adequately assess the status of the study device. Radiographs performed with the subject in a supine position.
Time Frame: 6 months and 12 months
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Study Arm (Dual Mobility) | Controlled Arm (Conventional)
Number analyzed (Participants) | 7 | 7
Participants
  6 months: number analyzed (Participants) | 4 | 3
  6 months: Yes | 0 | 0
  6 months: No | 4 | 3
  12 months: Yes | 0 | 0
  12 months: No | 7 | 7

ADVERSE EVENTS:
Time Frame: Adverse events collected upon device implantation to study termination, up to 12 months (±60 days)
Arm/Group | Study Arm (Dual Mobility) | Controlled Arm (Conventional)
All-Cause Mortality (participants affected / at risk) | 0/11 | 1/11
Serious Adverse Events (participants affected / at risk) | 3/11 | 3/11
Other Adverse Events (participants affected / at risk) | 3/11 | 4/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Arm (Dual Mobility) (N=11) | Controlled Arm (Conventional) (N=11)
RIGHTBUTTOCKBOIL (Skin and subcutaneous tissue disorders) | 1 | 0 — Not related to device or procedure
HYPOALBUMINEMIA (Blood and lymphatic system disorders) | 1 | 0 — Not related to device or procedure
HYDRONEPHROSIS WITH URETERAL STONES (Renal and urinary disorders) | 1 | 0 — Not related to device or procedure
HYPOHEMOGLOBIN (Blood and lymphatic system disorders) | 0 | 1 — Not related to device or procedure
RESPIRATORY BLEEDING (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Not related to device or procedure
BLURRED VISION IN THE LEFT EYE WITH DEFORMATION OF VISION FOR OVER SIX MONTHS (Eye disorders) | 0 | 1 — Not related to device or procedure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Arm (Dual Mobility) (N=11) | Controlled Arm (Conventional) (N=11)
COVID-19 IS POSITIVE (Infections and infestations) | 2 | 2 — Not related to device or procedure
LEFT CALF INTERMUSCULAR VEIN THROMBOSIS (Vascular disorders) | 0 | 1 — Not related to device or procedure
HYPOKALEMIA (Endocrine disorders) | 1 | 2 — Not related to device or procedure
HYPOALBUMINEMIA (Blood and lymphatic system disorders) | 1 | 1 — Not related to device or procedure

LIMITATIONS AND CAVEATS:
Only 22 participants were enrolled due to early termination of the study leading to a small number of participants analyzed for the outcome measures. No reliable conclusions could be made from the data collected and analyzed based on the small number of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-08-18): https://cdn.clinicaltrials.gov/large-docs/29/NCT04941729/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-29): https://cdn.clinicaltrials.gov/large-docs/29/NCT04941729/SAP_001.pdf